CLINICAL TRIAL: NCT06843018
Title: A Prospective, Open-label, Multicenter, Comparative, Randomised, Parallel-group Study to Evaluate the Efficacy and Safety of Different Doses of the Drug Graminidin With Anesthetic, a Metered Dose Topical Spray, in the Treatment of Acute Infectious and Inflammatory Pharyngeal Diseases Compared With Drug Septolete Total, Lozenges
Brief Title: Study to Evaluate the Efficacy and Safety of Different Doses of Graminidin With Anesthetic, a Metered Dose Topical Spray, in the Treatment of Acute Infectious and Inflammatory Pharyngeal Diseases Compared With Drug Septolete Total, Lozenges
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRM-02-06-2024
Record Dates: First submitted 2025-02-17; First posted 2025-02-24 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Pharyngitis Acute; Pharyngitis; Nasopharyngitis; Exacerbation of Chronic Pharyngitis
MeSH Terms: conditions — Pharyngitis; Nasopharyngitis | interventions — Anesthetics; benoxinate; Benzydamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Grammidin with anesthetic, 2 sprays every 6 hours (Experimental): Patients in group 1 will receive the drug Grammidin with anesthetic,a metered dose topical spray, with 2 sprays every 6 hours, three times a day under fed conditions for 7 days.
  Interventions: Drug: Grammidin with anesthetic
- Grammidin with anesthetic, 4 sprays every 6 hours (Experimental): Patients in group 2 will receive the drug Grammidin with anesthetic, a metered dose topical spray, with 4 sprays every 6 hours, three times a day under fed conditions for 7 days.
  Interventions: Drug: Grammidin with anesthetic
- Septolete Total, 1 lozenge every 6 hours (Active Comparator): Patients in group 3 will receive the drug Septolete Total, lozenges 3 mg + 1 mg, 1 lozenge every 6 hours, three times daily (maximum daily dose - 3 lozenges) for 7 days.
  Interventions: Drug: Septolete Total

INTERVENTIONS:
Drug: Grammidin with anesthetic — Grammidin with anesthetic, a metered dose topical spray
  Other Names: gramicidine C + oxybuprocaine + cetylpyridine chloride
  Arms: Grammidin with anesthetic, 2 sprays every 6 hours; Grammidin with anesthetic, 4 sprays every 6 hours
Drug: Septolete Total — Septolete Total, lozenges 3 mg + 1 mg
  Other Names: benzydamine + cetylpyridine chloride
  Arms: Septolete Total, 1 lozenge every 6 hours

SUMMARY:
This study aims to evaluete of tthe efficacy and safety of using different doses of the drug Grammidin with anesthetic, a metered dose topical spray, in the treatment of acute infectious and inflammatory pharyngeal diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 75 years inclusive.
2. Symptom "sore throat" due to infectious-inflammatory diseases of the pharynx (acute pharyngitis, acute nasopharyngitis, exacerbation of chronic pharyngitis) based on one or more of the following clinical manifestations:

   * Unpleasant sensations/discomfort in the throat - symptoms of pharyngeal paresthesia (scratchy throat, dryness or sore sensation ("foreign body" sensation));
   * Painful sensations in the throat, including sore throat at rest, throat burning, or pain upon swallowing saliva;
3. Severity of the symptom "sore throat" from 55 mm to 80 mm on the Visual Analog Scale (VAS).
4. A score of 5 to 8 points on the Clinical Symptom Severity Scale for tonsillopharyngitis.
5. Absence of indications for systemic antibacterial therapy at the time of inclusion in the study.
6. Negative test result for β-hemolytic streptococcus.
7. Duration of disease symptoms not exceeding 3 days at the time of inclusion in the study.
8. Women with a negative pregnancy test who have used one or more of the following contraceptive methods for 8 weeks prior to and during the 3 weeks after the end of the study: intrauterine devices (IUDs), oral contraceptives, contraceptive patches, long-acting injectable contraceptives, double barrier contraceptive method; or women who are infertile (documented conditions: hysterectomy, tubal ligation, infertility, menopause for more than 1 year); or men using a double barrier contraceptive method (condom with spermicide) throughout the study and for 3 weeks after its conclusion or men who are infertile (documented conditions: vasectomy, infertility).
9. Signed and dated informed consent form.

Non-inclusion Criteria:

1. Trauma and/or burns of the oropharynx, scarlet fever, rubella, measles at the time of inclusion in the study and not earlier than 3 months before inclusion in the study.
2. Treatment with any systemic antibacterial agents within 14 days prior to inclusion in the study.
3. Use of non-steroidal anti-inflammatory drugs and/or decongestants within 12 hours prior to the randomization visit.
4. Body temperature at screening and randomization visits ≥ 38.5 °C.
5. Infectious-inflammatory diseases requiring combined or systemic antibacterial therapy.
6. Severe, decompensated, or unstable somatic diseases (any diseases or conditions that threaten the patient's life or worsen the prognosis of the underlying disease, as well as make it impossible for the patient to participate in the clinical study).
7. History of malignancy, exept for subjects who have been disease-free for at least 5 years prior to screening.
8. Allergic history.
9. Participation in any other clinical study within 90 days prior to inclusion in the study.
10. Pregnancy or breastfeeding in women.
11. Refusal to use effective contraceptive methods during the study.
12. Alcoholism, drug addiction, abuse of psychotropic medications, including in history.
13. Smoking more than 10 cigarettes per day.
14. Positive urine test for narcotic substances and potent medications.
15. Vaccination within 21 days prior to study enrollment.
16. Other conditions that, in the opinion of the investigator, prevent the patient from being included in the study.

Exclusion Criteria:

1. Erroneous inclusion of a patient in the study (not meeting inclusion/exclusion criteria at the time of randomization).
2. Ineffectiveness of therapy. Therapy will be considered ineffective if there is no clinical improvement by Visit 2 (Day 3-4 of therapy) - persistence or worsening of the symptom "sore throat" and catarrhal phenomena compared to baseline data. If excluded, the patient will be assigned alternative treatment at the discretion of the investigator.
3. Patient non-compliance (a patient is considered compliant if the number of applications of the study drug/comparison drug is not less than 17 and not more than 25).
4. Smoking more than 10 cigarettes per day.
5. Requirement for prohibited concomitant therapy.
6. The investigator determines that continued participation in the study may pose a risk to the subject's safety or well-being.
7. Pregnancy or breastfeeding.
8. Gross violation by the patient of the study protocol procedures presented in the patient information sheet (PIS).
9. Withdrawal of informed consent (the patient's unwillingness to continue participation in the study).
10. Loss of contact with the patient (inability to reach the patient by mobile and home phone (if applicable), as well as through a contact person; there must be at least three documented attempts to contact the patient).
11. The emergence during the study of any diseases or conditions that worsen the patient's prognosis and make it impossible for the patient to continue participating in this clinical study.
12. Any other reasons, including administrative ones, that in the investigator's judgment would prevent the subject from completing the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Combined primary efficacy endpoint: VAS + TPA | Day 1 (Visit 1) - Day 8 (Visit 3)
  The primary efficacy endpoint will consist of two components:
  Change in sore throat severity as measured by the Visual Analog Scale (VAS) one hour after the first administration of the drug (STPID1h). In accordance to VAS, 0 mm - no pain, while 100 mm is the worst pain ever.
  Change in the severity of clinical symptoms according to the Tonsillopharyngitis Assessment Scale (TPA) at Visit 3 (or at the time of complete recovery and treatment completion if it occurs earlier). In accordance to TPA, each symptom is assessed from 0 points (absence or weak symptom) to 2 points (strong symptom).

SECONDARY OUTCOMES:
Change in sore throat severity, 30 min | Day 1 (Visit 1)
  Change in sore throat severity as measured by the Visual Analog Scale (VAS) 30 minutes after the first administration of the drug. In accordance to VAS, 0 mm - no pain, while 100 mm is the worst pain ever.
Change in sore throat severity, Visits 2 and 3 | Day 5 (Visit 2), Day 8 (Visit 3)
  Change in sore throat severity as measured by the VAS at Visits 2 and 3. In accordance to VAS, 0 mm - no pain, while 100 mm is the worst pain ever.
Change in the severity of clinical symptom | Day 5 (Visit 2)
  Change in the severity of clinical symptoms according to the Tonsillopharyngitis Assessment Scale at Visit 2. In accordance to TPA, each symptom is assessed from 0 points (absence or weak symptom) to 2 points (strong symptom).
Proportion of patients with no erythema and edema of the pharyngeal mucosa | Day 5 (Visit 2), Day 8 (Visit 3)
  Proportion of patients with no erythema and edema of the pharyngeal mucosa according to the Erythema and Edema subscale of the Tonsillopharyngitis Clinical Symptom Severity Scale at Visits 2 and 3.
Proportion of patients with no erythema and edema of the tonsils | Day 5 (Visit 2), Day 8 (Visit 3)
  Proportion of patients with no erythema and edema of the tonsils according to the Erythema and Edema subscale of the Tonsillopharyngitis Clinical Symptom Severity Scale at Visits 2 and 3.
Proportion of patients without signs of intoxication syndrome | Day 5 (Visit 2), Day 8 (Visit 3)
  Proportion of patients without signs of intoxication syndrome, assessed using a 4-point scale at Visits 2 and 3.
Overall frequency of adverse events | Screening, Day 1 (Visit 1) to Day 8 (Visit 3)
  Overall frequency of adverse events (AEs) (number of patients with at least one AE reported)
Number of adverse events | Screening, Day 1 (Visit 1) to Day 8 (Visit 3)
  Number of AEs stratified by severity and frequency
Frequency of drug-related adverse events | Day 1 (Visit 1) to Day 8 (Visit 3)
  Frequency of AEs related to the use of the study drug/comparison drug
Frequency of drug-related serious adverse events | Day 1 (Visit 1) to Day 8 (Visit 3)
  Frequency of serious adverse events (SAEs) related to the use of the study drug/comparison drug
Proportion of patients discontinued due to adverse events | Day 1 (Visit 1) to Day 8 (Visit 3)
  Proportion of patients who discontinued treatment due to AEs
Vital signs: systolic blood pressure | Screening, Day 1 (Visit 1), Day 5 (Visit 2), Day 8 (Visit 3)
  Systolic blood pressure (SBP, mmHg)
Vital signs: diastolic blood pressure | Screening, Day 1 (Visit 1), Day 5 (Visit 2), Day 8 (Visit 3)
  Diastolic blood pressure (DBP, mmHg)
Vital signs: heart rate | Screening, Day 1 (Visit 1), Day 5 (Visit 2), Day 8 (Visit 3)
  Heart rate (HR, bpm)
Vital signs: body temperature (Celsius temperature scale) | Screening, Day 1 (Visit 1), Day 5 (Visit 2), Day 8 (Visit 3)
  Body temperature (Celsius temperature scale)
Physical examination results: cardiovascular system | Screening, Day 1 (Visit 1), Day 5 (Visit 2), Day 8 (Visit 3)
  An assessment of the condition of the cardiovascular system on physical examination (normal condition or list of abnormal conditions, if any)
Physical examination results: respiratory system | Screening, Day 1 (Visit 1), Day 5 (Visit 2), Day 8 (Visit 3)
  An assessment of the condition of the respiratory system on physical examination (normal condition or list of abnormal conditions, if any)(normal condition or list of abnormal conditions, if any)
Physical examination results: digestive tract | Screening, Day 1 (Visit 1), Day 5 (Visit 2), Day 8 (Visit 3)
  An assessment of the condition of the digestive tract on physical examination (normal condition or list of abnormal conditions, if any)
Physical examination results: endocrine system | Screening, Day 1 (Visit 1), Day 5 (Visit 2), Day 8 (Visit 3)
  An assessment of the condition of the endocrine system on physical examination (normal condition or list of abnormal conditions, if any)
Physical examination results: musculoskeletal system | Screening, Day 1 (Visit 1), Day 5 (Visit 2), Day 8 (Visit 3)
  An assessment of the condition of the musculoskeletal system on physical examination (normal condition or list of abnormal conditions, if any)
Physical examination results: nervous system | Screening, Day 1 (Visit 1), Day 5 (Visit 2), Day 8 (Visit 3)
  An assessment of the condition of the nervous system on physical examination (normal condition or list of abnormal conditions, if any)
Physical examination results: sensory systems | Screening, Day 1 (Visit 1), Day 5 (Visit 2), Day 8 (Visit 3)
  An assessment of the condition of the sensory systems on physical examination (normal condition or list of abnormal conditions, if any)
Physical examination results: skin/visible mucous membranes | Screening, Day 1 (Visit 1), Day 5 (Visit 2), Day 8 (Visit 3)
  An assessment of the condition of the skin/visible mucous membranes on physical examination (normal condition or list of abnormal conditions, if any)
Results of laboratory and instrumental examinations: clinical blood test - hemoglobin | Screening, Day 8 (Visit 3)
  Hemoglobin (g/L)
Results of laboratory and instrumental examinations: clinical blood test - hematocrit | Screening, Day 8 (Visit 3)
  Hematocrit (%)
Results of laboratory and instrumental examinations: clinical blood test - red blood cell count | Screening, Day 8 (Visit 3)
  Red blood cell count (cells/L)
Results of laboratory and instrumental examinations: clinical blood test - platelet count | Screening, Day 8 (Visit 3)
  Platelet count (cells/L)
Results of laboratory and instrumental examinations: clinical blood test - leukocyte count | Screening, Day 8 (Visit 3)
  Leukocyte count (cells/L)
Results of laboratory and instrumental examinations: clinical blood test - erythrocyte sedimentation rate | Screening, Day 8 (Visit 3)
  Erythrocyte sedimentation rate (mm/h)
Results of laboratory and instrumental examinations: clinical blood test - myelocytes | Screening, Day 8 (Visit 3)
  Leukocyte formula (myelocytes, %)
Results of laboratory and instrumental examinations: clinical blood test - band neutrophils | Screening, Day 8 (Visit 3)
  Leukocyte formula (band neutrophils, %)
Results of laboratory and instrumental examinations: clinical blood test - segmented neutrophils | Screening, Day 8 (Visit 3)
  Leukocyte formula (segmented neutrophils, %)
Results of laboratory and instrumental examinations: clinical blood test - eosinophils | Screening, Day 8 (Visit 3)
  Leukocyte formula (eosinophils, %)
Results of laboratory and instrumental examinations: clinical blood test - basophils | Screening, Day 8 (Visit 3)
  Leukocyte formula (basophils, %)
Results of laboratory and instrumental examinations: clinical blood test - monocytes | Screening, Day 8 (Visit 3)
  Leukocyte formula (monocytes, %)
Results of laboratory and instrumental examinations: clinical blood test - lymphocytes | Screening, Day 8 (Visit 3)
  Leukocyte formula (lymphocytes, %)
Results of laboratory and instrumental examinations: blood chemistry - glucose | Screening, Day 8 (Visit 3)
  Glucose concentration (mmol/L)
Results of laboratory and instrumental examinations: blood chemistry - cholesterol | Screening, Day 8 (Visit 3)
  Total cholesterol concentration (mmol/L)
Results of laboratory and instrumental examinations: blood chemistry - protein | Screening, Day 8 (Visit 3)
  Total protein concentration (g/L)
Results of laboratory and instrumental examinations: blood chemistry - bilirubin | Screening, Day 8 (Visit 3)
  Total bilirubin concentration (micromol/L)
Results of laboratory and instrumental examinations: blood chemistry - creatinine | Screening, Day 8 (Visit 3)
  Creatinine concentration (micromol/L)
Results of laboratory and instrumental examinations: blood chemistry - alkaline phosphatase | Screening, Day 8 (Visit 3)
  Alkaline phosphatase activity (U/L)
Results of laboratory and instrumental examinations: blood chemistry - alanine transaminase | Screening, Day 8 (Visit 3)
  Alanine transaminase activity (U/L)
Results of laboratory and instrumental examinations: blood chemistry - aspartate transaminase | Screening, Day 8 (Visit 3)
  Aspartate transaminase activity (U/L)
Results of laboratory and instrumental examinations: urinalysis - specific gravity | Screening, Day 8 (Visit 3)
  Specific gravity of the urine
Results of laboratory and instrumental examinations: urinalysis - pH | Screening, Day 8 (Visit 3)
  pH of the urine
Results of laboratory and instrumental examinations: urinalysis - protein | Screening, Day 8 (Visit 3)
  Protein concentration (g/L)
Results of laboratory and instrumental examinations: urinalysis - glucose | Screening, Day 8 (Visit 3)
  Glucose concentration (mmol/L)
Results of laboratory and instrumental examinations: urinalysis - red blood cells | Screening, Day 8 (Visit 3)
  Red blood cell content (number in sight)
Results of laboratory and instrumental examinations: urinalysis - white blood cells | Screening, Day 8 (Visit 3)
  White blood cell content (number in sight)
Results of laboratory and instrumental examinations: blood chemistry - glomerular filtration rate | Screening, Day 8 (Visit 3)
  Glomerular filtration rate calculated using blood creatinine levels and formula CKD-EPI

CONTACTS AND LOCATIONS:
Locations (12):
- Russia (12):
  - State autonomous health care institution "Engels City Clinical Hospital No. 1", Engel's
  - State Budgetary Healthcare Institution of the Kaliningrad Region "City Hospital No. 2.", Kaliningrad
  - Unimed-C Jsc, Moscow
  - Professors' Clinic LLC., Perm
  - Limited Liability Company "Medical Center Eco-Safety", Saint Petersburg
  - Aurora MedFort LLC, Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Polyclinic No. 117", Saint Petersburg
  - Limited Liability Company "Clinic Zvezdnaya", Saint Petersburg
  - Limited Liability Company "Meili", Saint Petersburg
  - LLC "Mariel Clinic", Saint Petersburg
  - LLC "Center for DNA Research", Saratov
  - LLC "Polyclinic Polimedika Veliky Novgorod", Veliky Novgorod

IPD SHARING:
Plan to Share IPD: No